CLINICAL TRIAL: NCT05345626
Title: It is Possible to Continuous Monitor Vital Signs in Patients Discharged a Rehabilitation Center - An Observational Feasibility Study
Brief Title: Vital Signs Monitoring in Rehabilitation Center Patients
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Eske Kvanner Aasvang, Professor, Rigshospitalet, Denmark
Other Study IDs: Rigshospitalet, Copenhagen
Record Dates: First submitted 2022-04-12; First posted 2022-04-26 (Actual); Last update posted 2022-05-13 (Actual); Status verified 2022-05

CONDITIONS: Comorbidities
Keywords: Rehabilitation patients, wireless monitoring, vital signs

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Some patients unable to return home from hospital due to physical or mental illness will be discharged to a rehabilitation home to restore strength and rehabilitate. This study attempts to examine if it is possible to continuously monitor the vital signs in patients discharged to a rehabilitation center and whether wearable devices will detect more abnormal vital signs than the rehabilitation facility, as well as complication and readmission rates.

DETAILED DESCRIPTION:
Patients who are ready to leave the hospital but are deemed unable to return home are discharged to a rehabilitation center to regain strength and performance.

Vital signs are only measured when deemed necessary at the rehabilitation center, in contrast to hospital wards, where vital signs are measured intermittently and manually every 8-12 hours.

Wearable devices that continuously monitor a patient's vital signs may be able to detect patients who are deteriorating, as abnormal vital signs often precede a physiologic decline This study aims to determine whether it is possible to continuously monitor patients discharged to a rehabilitation center and detect more abnormal vital signs than measurements from the rehabilitation center. By attaching three wearable devices to 20 patients, we wished to record the vital signs for up to 96 hours, documenting abnormal vital signs as well as complications - and readmission rates.

ELIGIBILITY:
Inclusion Criteria:

* discharged to the rehabilitation center after surgery or; diagnosed with ischemic heart disease, chronic heart disease, apoplexia cerebri, chronic obstructive pulmonary disease, or diabetes.
* Inclusion less than 72 h from rehabilitation admission

Exclusion Criteria:

* Unable to give informed consent
* Implanted pacemaker or cardioverter-defibrillator
* allergic to plaster, plastic, silicone

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospital patients discharged to a rehabilitation center
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2019-10-14 (Actual); Primary Completion 2021-09-08 (Actual); Study Completion 2021-10-08 (Actual)

PRIMARY OUTCOMES:
Monitoring time | 96 hours
  Monitoring time with data from any device

SECONDARY OUTCOMES:
SpO2 < 92% | 96 hours
  Duration of SpO2 < 92%
SpO2 < 88% | 96 hours
  Duration of SpO2 < 88%
SpO2 < 85% | 96 hours
  Duration of SpO2 < 85%
SpO2 < 80% | 96 hours
  Duration of SpO2 < 80%
Respiratory rate <5 breaths per minute | 96 hours
  Duration of respiratory rate <5 breaths per minute
Respiratory rate <11 breaths per minute | 96 hours
  Duration of respiratory rate <11 breaths per minute
Respiratory rate >24 breaths per minute | 96 hours
  Duration of respiratory rate >24 breaths per minute
Respiratory rate >30 breaths per minute | 96 hours
  Duration of respiratory rate >30 breaths per minute
Heart rate <30 beats per minute | 96 hours
  Duration of heart rate <30 beats per minute
Heart rate <40 beats per minute | 96 hours
  Duration of heart rate <40 beats per minute
Heart rate > 110 beats per minute | 96 hours
  Duration of heart rate > 110 beats per minute
Heart rate > 130 beats per minute | 96 hours
  Duration of heart rate > 130 beats per minute
Systolic blood pressure <70 mmHg | 96 hours
  Number of systolic blood pressure <70 mmHg measurements
Systolic blood pressure <90 mmHg | 96 hours
  Number of systolic blood pressure <90 mmHg measurements
Systolic blood pressure >180 mmHg | 96 hours
  Number of systolic blood pressure >180 mmHg measurements
Systolic blood pressure >220 mmHg | 96 hours
  Number of systolic blood pressure >220 mmHg measurements

OTHER OUTCOMES:
Complication | 30 days
  Complication frequency within 30 days from study inclusion
Readmission | 30 days
  Readmission frequency within 30 days from study inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Eske K Aasvang, Dr. Med, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Center for Rehabilitering og Akutpleje - Bystævneparken, Brønshøj, Denmark

IPD SHARING:
Plan to Share IPD: Undecided